CLINICAL TRIAL: NCT04912414
Title: Brief Family Therapy (BFT) for the Treatment of Psychosomatic Symptoms in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Responsible Party: Principal Investigator, Francoise Uwizeye, Principal investigator, University of Rwanda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017/CMHS IRB/2020
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Patient Engagement
Keywords: Psychosomatic symptom; Anxiety; Brief Family Therapy; Session
MeSH Terms: conditions — Patient Participation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Family Therapy (BFT) for the treatment of psychosomatic symptoms in Rwanda (Experimental): The participants from the control group were assigned to the Brief Family Therapy for reducing the medically unexplained symptoms. But the control group was not assigned to the intervention (BFT).
  Interventions: Behavioral: Brief Family Therapy (BFT)

INTERVENTIONS:
Behavioral: Brief Family Therapy (BFT) — Patients transferred to the hospital for the treatment of psychosomatic symptoms was randomized (1:1) to receive either Brief Family Therapy (BFT) or a control treatment. Some participants randomized to the BFT arm receive a combination of chemotherapy and BFT and others receive only BFT. BFT comprises 10 sessions using a generic model of problem formation and resolution. This psychotherapy is useful for treating individual, couple, and family problems. Its broad applicability is based on its view that the client's complaint is the problem, not a symptom of something else BFT views behavior, especially a client's problematic behavior, as a function of interaction with other people. After randomization, all participants were asked to complete questionnaires about their psychosomatic symptoms and health at baseline, at the end of the intervention (at 4 months).

SUMMARY:
Mental health is fundamental part of the human being worldwide taken as the driver of all daily activities of the people. Psychosomatic disorders are the psychological diseases that are the burden in mental health worldwide. These diseases characterized by the medically unexplained symptomatology (MUS) are considered as a comprehensive, interdisciplinary framework for assessment of psychological factors affecting individual vulnerability, as well as course and outcome of illness; biopsychosocial consideration of patient care in clinical practice; specialist interventions to integrate psychological therapies in the prevention, treatment, and rehabilitation of medical disease. This psychosomatic symptomatology is highly prevalent in developing countries. Prior studies stated that Brief family therapy (BFT) is an effective for MUS. Some possible reasons could be solving conflicts and interpersonal problems by means of training certain skills such as problem solving, developing relationships with others, effective coping, assertiveness and positive thinking. This quasi-experimental design investigates whether BFT can reduce psychosomatic symptoms in Kibungo referral hospital of Eastern Province, Rwanda. Experimental group enroll 60 patients who will be followed up during 2 months. Control group enroll 60 patients. Participants from experimental group will attend 8 sessions of BFT. Statistical analyses will be performed using the SPSS software version 22. As recommended by the declaration of Helsinki, confidentiality and voluntariness were ensured. Informed consents were obtained from the participants. Paired-samples t-test will be used for assessing the means differences between two groups before and after the BFT. 95% of confidence intervals and 5% of statistical significance are applied. In the baseline, sociodemographic questionnaire and psychometric tools will be provided. The psychometric tools will be used in the baseline and at the end of BFT sessions.

DETAILED DESCRIPTION:
Background and study aims Medically unexplained symptoms (MUS) is a diagnosis given to people with long-term physical problems that do not match any recognised medical conditions. Psychosomatic symptoms are physical problems such as pain that are a result of- or made worse by- emotional stress or depression. In some cases, the body's immune system may be weakened by severe and/or chronic stress. Psychosomatic symptoms are common and can greatly impact quality of life. There are not many treatments for psychosomatic symptoms, and treatment of these symptoms are not prioritized as their cause is unexplained by modern medicine.

Aim of the study This study aims to investigate whether a brief family therapy program can reduce psychosomatic symptoms in Kibungo referral hospital of Eastern Province, Rwanda.

Who can participate? Adults diagnosed with medically unexplained symptoms (MUS) What does the study involve? Patients transferred to the participating centre for the treatment of psychosomatic symptoms were treated with either Brief Family Therapy (BFT) or a control treatment for 2 months.

Participants were allocated to one of the two groups, with an equal chance of being in either group. At the start of the study, all participants were provided with questionnaires for assessing their baseline characteristics and their expectations about the treatment. The participants were also be asked to complete questionnaires about their psychosomatic symptoms and health at the start and at the end of the study. What are the possible benefits and risks of participating? The benefits of participating were psychological support provided by BFT. Benefits will be explained to participants and then provided the consent form for participating in the research.

They were also promised that they could withdraw at any time and no asked any reason about their participation. Privacy and confidentiality were respected in this study for protecting participants. No risks are anticipated from participation in this study.

Where is the study run from? The study run from University of Rwanda (Rwanda) and was conducted in the medical setting.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-59 years
* Being diagnosed Medically Unexplained Symptoms at least more than once with the similar symptoms.
* Being with psychosomatic at least more than 6 months

Exclusion Criteria:

* Having no will to participate in the study;
* Not signing the informed consents to participate

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Psychosomatic Symptom Checklist (PSC-17) | Two months or eight weeks of the follow-up
  Psychosomatic Symptom Checklist (PSC-17) is psychometric instrument used to assess the psychosomatic symptoms among the patients seeking health care at the health setting. Paired-sample t-test was used to assess how an BFT contributed to a reduction of psychosomatic symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Uwizeye, Mr., Principal Investigator — University of Rwanda
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
As the data was collected from the patients and they were collected anonymously, the data may be shared with other researchers when request.